CLINICAL TRIAL: NCT01854385
Title: Sumatriptan as Treatment for Moderate to Severe Post-Traumatic Headache
Brief Title: Sumatriptan as Treatment for Post-traumatic Headache
Acronym: TWIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jeanne Hoffman, Professor- Rehabilitative Medicine: Psychology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 44912
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Post-traumatic Headache
Keywords: Post-traumatic headache; Traumatic brain injury; Sumatriptan
MeSH Terms: conditions — Post-Traumatic Headache; Brain Injuries, Traumatic | interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sumatriptan (Experimental): Open label study of sumatriptan to treat post-traumatic headache. Subjects will use sumatriptan 100 mg at the onset of headache pain and may repeat the dose if not pain-free in 2 hours. Subjects will receive a maximum of 18 pills for use over two months. Subjects will maintain a daily headache diary.
  Interventions: Drug: Sumatriptan 100 mg

INTERVENTIONS:
Drug: Sumatriptan 100 mg — This is a single-arm, unblinded study of treatment for post-traumatic headache with the open label medication sumatriptan and is being undertaken to test necessary study instruments and procedures, establish feasibility and determine side effects in a population with complicated mild, moderate and severe TBI.
  Other Names: Imitrex; Imigran

SUMMARY:
This phase II evaluation of sumatriptan as a treatment for post traumatic headache (PTH) will examine the methods and approach necessary to take the next step to a phase III trial. The sample will include 40 persons with mild complicated, moderate or severe TBI who will be recruited from patients discharged from the acute rehabilitation unit as well as outpatient clinics and the community who are between 3 and 24 months of injury and will be followed over 3 months. The investigators plan to enroll those who have moderate to severe headache with frequency of at least four and up to a maximum of fifteen total headache days per month and at least three months after discharge from hospital. The investigators will use headache diaries to track the headaches for a month. If subjects still have significant headache, the investigators will instruct them in the use of sumatriptan 100 mg. to treat headaches. The subjects will continue to keep daily headache diaries. The investigators will evaluate them at baseline, Day 30 and Day 90. Each subject will receive weekly telephone follow up calls from the research staff. The investigators will measure pain severity, duration, recurrence of headaches, and side effects and how well persons with TBI can use headache diaries.

DETAILED DESCRIPTION:
I. Specific Aims of Study: The ultimate aim of this Phase II open-label study is to test the research methods and approach necessary to successfully carry out a Phase III study for the treatment of post-traumatic headache (PTH). During this study, we will

1. Determine the feasibility of using a headache diary accessed via smart phone application, the web, or paper/pencil to record accurate headache data in a group of individuals with TBI, and their caregivers as indicated.
2. Evaluate the approximate effect size of sumatriptan on pain severity, duration, and recurrence of headaches in persons with moderate to severe PTH in order to establish the necessary sample size for a Phase III study.
3. Assess the side effect profile of sumatriptan in a brain-injured population as well as the safety of sumatriptan in subjects with TBI.
4. Evaluate the ability of persons with TBI, and their caregivers as indicated, to successfully use abortive headache medications and comply with treatment.
5. Examine the relationship between PTH and cognitive, emotional, and other self-report measures to determine important factors to include in a Phase III study.

This is a single arm, unblinded study enrolling 40 subjects and is being undertaken to test necessary study instruments and procedures, establish feasibility and determine side effects in a population with mild complicated, moderate or severe TBI in preparation for a subsequent Phase III study.

Data collection will occur at enrollment (Clinic Visit 1) at which baseline testing will occur, Day 30 (Clinic Visit 2), and Day 90 (Clinic Visit 3).

Pre-treatment Visit (Visit 1): Subjects who complete informed consent and meet the inclusion criteria (with no exclusion criteria) will be asked to complete 30 days of headache diary to document the number of headaches, headache severity, headache days and description of their headache and associated symptoms. Research staff will contact them on a weekly basis to answer questions and maximize accuracy and compliance with the diary. Proper utilization of a headache diary and success of data input by the subject and caregiver will be evaluated following weekly interviews with the research assistant.

Treatment Visit (Clinic Visit 2):

A medical history will be obtained to review inclusion and exclusion criteria and to elicit a thorough review of systems so that adverse events will be identifiable if they occur. Physical examination will also ensure that cardiovascular status is compatible with sumatriptan use and will document current status to allow for identification of potential adverse events. Finally, standard primary headache classification criteria will be reviewed with each patient to determine whether they meet criteria for migraine or probable migraine. Headache histories will be assessed and subjects that have experienced between 4-15 headaches will be included in the medication intervention with Sumatriptan. Subjects who qualify for the Sumatriptan intervention will receive several assessments, given medication, usage instructions, and scheduled for weekly phone calls for weeks 5-11. Individuals whose headaches do not meet criteria for migraine or probable migraine, based on data from headache diaries, will have their participation in the study end.

Weekly Telephone Follow-Up Calls: Research staff will call each participant weekly to check on compliance with drug diary use during the first month of the study (Weekly calls 1-3) to check on compliance in diary usage. For weekly calls in weeks 5-11 (for the intervention participants), research staff will inquire about study drug usage, and query for adverse events. Use of rescue medications for headache will be recorded. In the case of minor adverse effects which are bothersome to the patient, the dosage will be decreased by ½ pill per use.

Follow up Visit (Visit 3). This will be the final visit for the subjects. Vital signs will be obtained. Drug containers and headache diaries will be collected from all subjects. Outcome measures will be administered.

Use of sumatriptan and rescue drug: Two packages of nine (9) sumatriptan 100- mg. pills (18 pills total for 2 months of treatment) will be dispensed to each subject on Day 30 once they have gone through baseline assessment. On average, this will treat a minimum of 5 headaches or a maximum of 9 headaches per month. Subjects will be instructed to take the sumatriptan at the onset of headache pain. If subjects are not pain free at 2 hours after the first dose of study medication, they will be allowed to take one additional pill, but will be limited to 2 pills in a 24 hour period. Subjects will be instructed to take no more than 9 pills in a 30 day period based on research which suggests that additional dosages may increase the risk of medication-overuse headache. A list of appropriate medications will be provided that they can use if they: 1) continue to have headache pain 2 hours after their second dose of study drug, or 2) they have used their 30 day supply of study drug within the month. All subjects will be contacted by telephone on a weekly basis to review their headache diaries, assess potential adverse events, review compliance with use of the study drug, assess other treatments being utilized, and answer any questions.

Data Analysis: Data analysis for the feasibility and safety aims will be primarily descriptive. The investigators will calculate the percent of subjects who used the diary successfully, percent who stopped taking sumatriptan because of side effects, percent who experienced each adverse event, and percent who were able to maintain compliance with treatment. A confidence interval will be determined for each estimate. To get preliminary data on efficacy of sumatriptan, headache control will be compared before and after the participants start taking sumatriptan. The investigators will calculate the percent of headaches that had complete resolution (pain free at 2 hours) for each person, during the initial (pre-intervention) month when they used their regular treatment and during the two months (intervention) when they treated headaches with sumatriptan and compare them using a paired t-test. The investigators will also examine different definitions of headache relief (pain free by 30 minutes, no more than mild pain (score <=1) by 30 minutes, no more than mild pain by 2 hours) to see if another outcome measure may have advantages for a future Phase III study. Any differences in compliance, side effects, and feasibility based on cognitive functioning will be described, as well as by other self-report and emotional health measures. Changes in these measures from pre to post treatment will also be examined to determine whether there is any change that occurs with treatment and which may be important variables to include in a Phase III study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65. The lower age limit is set for ability to consent as an adult for research participation as well as being a minimum age for administration of most validated outcome measurements. The higher age limit is set to 65 to reduce likelihood of health issues which may be a contraindication to the use of sumatriptan and to meet recommendations by the International Headache Society.62
* Diagnosis of TBI occurring at least 3 months but not greater than 60 months before enrollment. Three months was chosen to include only those subjects who are having headache beyond their acute injury and 60 months to identify the ability of individuals with TBI and headache to use both a headache diary and the medication.
* Subject has at least four and up to a maximum of fifteen total headache days per month. Subject report of meeting this criteria will result in the subject entering the first month of the study. However, this frequency must be documented in headache diary to enter the treatment phase of the study.
* Headaches are classified as moderate to severe (2 or 3 on the 4 point pain scale: 0=no headache, 1=mild headache, 2=moderate headache, 3=severe headache). As above, headache severity must be documented in the month-long headache diary prior to entry into the treatment phase.
* Subject is able and willing to give written informed consent for participation in screening activities and to participate fully in the study if eligible. For those subjects who score below 25 on the Mini Mental Status Examination, there must be a caregiver willing to also be consented for participation in the study.
* Female subjects of childbearing potential must have a negative pregnancy test at enrollment, and agree to remain abstinent or use acceptable methods of birth control (i.e., hormonal contraceptives, intrauterine device, diaphragm with spermicide, cervical cap or sponge, condoms, or partner has had a vasectomy). Sumatriptan has been assigned to pregnancy category C by the FDA. Animal studies have revealed evidence of decreased fetal body weight, embryo lethality, and cervicothoracic vascular defects. There are no controlled data in human pregnancy and therefore, sumatriptan should only be given during pregnancy when benefit outweighs risk.

Exclusion Criteria:

* History of ischemic heart disease (angina pectoris, history of myocardial infarction, silent ischemia, Prinzmetal's angina/coronary vasospasm, ischemic bowel disease, or peripheral vascular disease) based on self-report or history of basilar or hemiplegic migraine.
* Uncontrolled hypertension at initial visit (sitting systolic pressure > 140 mm Hg, diastolic pressure > 90 mm Hg).
* Impaired renal or liver function by medical history.
* Subject has taken an MAO inhibitor within 2 weeks of screening because these drugs and sumatriptan use the same metabolic pathway.
* Subject has hypersensitivity reactions or other intolerance to sumatriptan or any other 5-HT 1B/1D-receptor agonists.
* If subjects have medication overuse headache in the opinion of the investigator (if using medication to treat acute headache on more than 15 days per month).
* Inability to speak or read English which would limit ability to interact with examiners and complete headache diary and other questionnaires during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M Hoffman, PhD, Principal Investigator — University of Washington; Leslie Kempthorne, Study Director — University of Washington
Locations (2):
- United States (2):
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma TL, Lucas S, Barber J, Hoffman JM. Pilot study evaluating treatment with sumatriptan for moderate to severe post-traumatic headache: A phase 2 open-label study. Headache. 2024 Oct;64(9):1135-1142. doi: 10.1111/head.14807. Epub 2024 Aug 13. PMID 39136260
- See also: University of Washington TBI Model System — https://tbi.washington.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between August 2013 and January 2018.
Period: Pre-Treatment
Arm/Group | Sumatriptan
Started | 40
Completed | 17
Not Completed | 23
Not completed — Withdrawal by Subject | 4
Not completed — Did not meet criteria based on headache number | 15
Not completed — Disqualified based on blood pressure requirement | 3
Not completed — Unable to come for study visits | 1
Period: Treatment
Arm/Group | Sumatriptan
Started | 17
Completed | 16
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sumatriptan
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 27
  Race: Black | 3
  Race: Asian/Pacific Islander | 3
  Race: Hispanic | 5
  Race: Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 40
Post-Injury Months [Mean (Standard Deviation); unit: months] — Population: Exact injury date unknown for two participants.
  months
    number analyzed (Participants) | 38
    (all) | 13.4 (11.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Headache Relief
Description: percent of headaches that had complete resolution (pain free at 2 hours) for each person, during the initial (pre-intervention) month when they used their regular treatment and during the second of the two months (intervention) when they treated headaches with sumatriptan compared using a mixed-effects regression model. Reported number is the difference in headache resolution from the pre-intervention headaches to the intervention headaches.
Time Frame: 1 month
Population: Subjects with complete pre-intervention and intervention data
Measure: Mean (95% Confidence Interval); unit: percentage of headaches resolved
Arm/Group | Sumatriptan
Number analyzed (Participants) | 11
percentage of headaches resolved | 23 [-3 to 50]
Statistical Analysis 1: Comparison: Sumatriptan; Test type: Superiority; p = .079, Mixed Models Analysis

2. Secondary Outcome: Adverse Events
Description: The investigators will calculate the percent who stopped taking sumatriptan because of side effects, percent who experienced each adverse event.
Time Frame: 2 months
Population: participants that completed the intervention
Measure: Number; unit: participants
Arm/Group | Sumatriptan
Number analyzed (Participants) | 15
participants
  Stopped taking sumatriptan due to side effects | 0
  Rebound headaches | 1
  Fatigue/drowsiness | 2
  Dizziness | 2
  Gastrointestinal symptoms | 4
  Numbness/Tingling | 2
  Itch/rash | 1
  Joint pain | 1
  Restlessness | 1
  Sweating/flushing | 2
  Elevated blood pressure | 1
  Anxiety | 1
  Sore Throat | 1

3. Secondary Outcome: Headache Diary Compliance
Description: The investigators will calculate the mean percentage of headache diary completion of intervention subjects in the final month of participation.
Time Frame: 1 month
Population: participants that completed the intervention with valid diary entries
Measure: Mean (Standard Deviation); unit: percentage of diary days completed
Arm/Group | Sumatriptan
Number analyzed (Participants) | 15
percentage of diary days completed | 80 (22)

4. Secondary Outcome: Sumatriptan Compliance
Description: Mean rate of headaches treated with sumatriptan in final month of intervention.
Time Frame: 1 month
Population: participants that completed the intervention with valid diary entries
Measure: Mean (Standard Deviation); unit: percentage of headaches
Arm/Group | Sumatriptan
Number analyzed (Participants) | 15
percentage of headaches | 25 (22)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from participants who enrolled in the intervention portion of the study, from the time of consent and dispensation of study drug until the end of their study treatment follow-up - approximately three months. For this study, the end of the study treatment follow-up is defined as 30 days following the last study clinic visit.
Arm/Group | Sumatriptan
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 9/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sumatriptan (N=17)
Rebound headaches (Nervous system disorders) | 1 (1)
Fatigue/Drowsiness (Nervous system disorders) | 2 (5)
Dizziness (Nervous system disorders) | 2 (2)
Gastrointestinal Issues (Gastrointestinal disorders) | 4 (6) — nausea, upset stomach, intestinal discomfort, esophageal discomfort
Numbness/Tingling (General disorders) | 2 (2)
Itch/Rash (General disorders) | 1 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Restlessness (Nervous system disorders) | 1 (2)
Sweating/Flushing (Vascular disorders) | 2 (5)
Elevated blood pressure (Vascular disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT01854385/Prot_SAP_001.pdf